CLINICAL TRIAL: NCT02156011
Title: Kinematics and Joint Loading in Total Knee Arthroplasty
Brief Title: Comprehensive Assessment of the Musculoskeletal System
Acronym: CAMS-Knee
Status: Completed | Type: Observational
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Robert Mathys Stiftung, Bettlach, Switzerland (Unknown); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, William R. Taylor, Professor of Movement Biomechanics, Swiss Federal Institute of Technology
Other Study IDs: EK 2013-N-90; EA4/069/06 (Other: Charite-Universitätsmedizin Berlin Germany)
Record Dates: First submitted 2014-06-02; First posted 2014-06-05 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Total Knee Arthroplasty
Keywords: In vivo knee joint kinematics; In vivo knee joint loading; Video-fluoroscopy; Instrumented implants; Optical motion capture; Ground reaction forces; Electromyography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Instrumented knee implant: 4-6 subjects with an instrumented TKA, that has been implanted within the study "Kniemessprothese: Belastungsmessung bei Patienten mittels einer instrumentierten Knie-Endoprothese" (EA4/069/06) approved and conducted at the Charité- Universitätsmedizin in Berlin, Germany, will be involved in this project.

SUMMARY:
The objective of this research is to synchronously assess in vivo loading data of the knee joint, tibio-femoral 3D kinematics by means of automated video-fluoroscopy, whole leg kinematics by means of skin markers, ground reaction forces, as well as muscle activity patterns in 4 to 6 subjects with instrumented total knee arthroplasty (TKA) during dynamic functional activities of daily life. The comprehensive in vivo dataset will provide unique information to evaluate the relationship between the kinematics, respectively the alignment of the TKA, and the resulting loading of the implant in vivo.

The whole data package will be made available for download on a public database, such that it can be utilized for the testing and improvement of TKA designs as well as for the validation and improvement of musculoskeletal modelling by researchers around the world.

DETAILED DESCRIPTION:
STUDY SUBJECTS:

4-6 subjects with an instrumented TKA, that has been implanted within the study "Kniemessprothese: Belastungsmessung bei Patienten mittels einer instrumentierten Knie-Endoprothese" (EA4/069/06) approved and conducted at the Charité- Universitätsmedizin in Berlin, Germany, will be involved in this project. This instrumented prosthesis was implanted in 9 subjects with osteoarthritis.

DATA ACQUISITION:

The testing will be performed at the Institute for Biomechanics at the ETH Zurich. The kinematic and kinetic measurements include video-fluoroscopic tibio-femoral 3D implant motion; whole leg motion capture based on skin markers as well as ground reaction forces. Simultaneously the joint loading is assessed by means of the instrumented TKA and a telemetry unit for transmitting the strain gage signals. In all subjects, muscle activity is additionally simultaneously assessed using surface electromyography (EMG). The electrodes are placed onto the skin at the sites of eight muscles in the lower limbs. At the beginning of the test session, the maximal voluntary contraction will be assessed by means of the EMG electrodes, performing the following four motion tasks:

* One legged standing and lifting the heel to stand on tiptoe.
* Extension of the knee joint against a load by means of a strap around the lower leg just above the ankle. (Subject is sitting on a bench, lower legs are hanging down).
* Flexion of the knee joint against a load by means of a strap around the lower leg just above the ankle. (Subject is sitting on a bench, lower legs are hanging down).
* Dorsiflexion of the ankle against a manual resistant force of the investigator. (Subject is sitting on a bench, lower legs are hanging down).

To familiarize the subjects with the dynamic data acquisition protocol, six test trials will be conducted that just include the motion capture system (motion capture trials, each performed twice). This is followed by the main test procedure, which will consist of two static (static trials) and three dynamic trials (dynamic trials) assessed simultaneously by the video-fluoroscopy, the motion capture systems the force plates, as well as the instrumented TKA. During the dynamic trials the fluoroscopic measurement unit mounted on an automated trolley will move along the subject and capture the motion of the knee in question.

Motion capture trials:

* Standing trial in an anatomic upright position
* Calibration motion (Standing in upright position, followed by free movement of legs and arms)
* Four basic motion tasks to define functional estimated joint axis, respectively centers: dorsiplantarflexion motion of the ankle, inversion/eversion motion of the ankle, flexion/extension motion of the knee, hip circumduction (List et al., 2012b)

Static trials:

* Standing trial in an anatomic upright position captured from the side.
* Standing trial in an anatomic upright position captured from an angle of 45°.

Dynamic trials:

For each of the following activities the subjects has to perform five valid gait cycles or repetitions respectively. A trial is considered valid, when the knee is in the field of view of the image intensifier during the whole cycle and the force plate got hit for level gait, walking downhill and stair descent.

* Level gait
* Stair descent a two steps staircase
* Downhill walking a 10° inclined slope
* Sit down and stand up from a chair
* Squatting

For documentation, all dynamic trials will additionally be captured by two video cameras. All anonymized data will be made available for download on a public database.

ELIGIBILITY:
Inclusion Criteria:

* Instrumented TKA
* Participant of the study EA4/069/06, Charité- Universitätsmedizin Berlin, Germany,

Exclusion Criteria:

* Not able to walk freely without walking aid
* Any medical condition that could impact on study results

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after total knee replacement surgery from the Charité- Universitätsmedizin in Berlin, Germany
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2017-10-09 (Actual)

PRIMARY OUTCOMES:
Video-fluoroscopy outcome parameters (kinematic parameters): | up to 4 weeks
  Quantification of the 3D kinematics of the TKA knee through fitting subject-specific 3D computer aided design models to the video-fluoroscopic data during functional activities.
Knee joint loading outcome parameters (kinetic parameters) | up to 4 weeks
  In vivo measurements of internal joint contact forces and moments through the use of instrumented implants that are capable of non-invasively transmitting the forces and moments measured within the joint.

SECONDARY OUTCOMES:
Optical motion capture outcome parameters | up to 4 weeks
  By means of optical motion capture with passive reflective skin markers, the 3D motion patterns of the entire ipsi- as well as contralateral lower limbs is assessed. This allows the identification of left-right asymmetries and compensation motion in adjacent joints and/or joints of the contralateral leg.
Ground reaction force outcome parameters: | up to 4 weeks
  The simultaneous measurements of ground reaction forces during dynamic activities allows the assessment of time/distance gait parameters as well as the identification of limping in individual patients
Electromyography outcome parameters | up to 4 weeks
  In all subjects muscle activity during functional activity is additionally simultaneously assessed using surface electromyography (EMG). The electrodes are placed onto the skin at the sites of eight muscles in the lower limbs.

OTHER OUTCOMES:
Clinical outcome parameters | already available
  * Radiographically assessed alignment
  * Actual pain intensity measured with Visual Analog Scale (VAS)
  * WOMAC, KSS score, Forgotten Joint Score

CONTACTS AND LOCATIONS:
Overall Officials: William R Taylor, PhD, Principal Investigator — Institute for Biomechanics ETH Zurich Switzerland
Locations (1):
- Institute for Biomechanics, ETH Zurich, Zurich, Switzerland

REFERENCES:
- [Background] Konig C, Sharenkov A, Matziolis G, Taylor WR, Perka C, Duda GN, Heller MO. Joint line elevation in revision TKA leads to increased patellofemoral contact forces. J Orthop Res. 2010 Jan;28(1):1-5. doi: 10.1002/jor.20952. PMID 19637213
- [Background] Konig C, Matziolis G, Sharenkov A, Taylor WR, Perka C, Duda GN, Heller MO. Collateral ligament length change patterns after joint line elevation may not explain midflexion instability following TKA. Med Eng Phys. 2011 Dec;33(10):1303-8. doi: 10.1016/j.medengphy.2011.06.008. Epub 2011 Jul 20. PMID 21764353
- [Background] Taylor WR, Heller MO, Bergmann G, Duda GN. Tibio-femoral loading during human gait and stair climbing. J Orthop Res. 2004 May;22(3):625-32. doi: 10.1016/j.orthres.2003.09.003. PMID 15099644
- [Background] Trepczynski A, Kutzner I, Kornaropoulos E, Taylor WR, Duda GN, Bergmann G, Heller MO. Patellofemoral joint contact forces during activities with high knee flexion. J Orthop Res. 2012 Mar;30(3):408-15. doi: 10.1002/jor.21540. Epub 2011 Aug 30. PMID 22267190
- [Background] Zihlmann MS, Gerber H, Stacoff A, Burckhardt K, Szekely G, Stussi E. Three-dimensional kinematics and kinetics of total knee arthroplasty during level walking using single plane video-fluoroscopy and force plates: a pilot study. Gait Posture. 2006 Dec;24(4):475-81. doi: 10.1016/j.gaitpost.2005.12.012. Epub 2006 Feb 10. PMID 16473011
- [Background] List R, Foresti M, Gerber H, Goldhahn J, Rippstein P, Stussi E. Three-dimensional kinematics of an unconstrained ankle arthroplasty: a preliminary in vivo videofluoroscopic feasibility study. Foot Ankle Int. 2012 Oct;33(10):883-92. doi: 10.3113/FAI.2012.0883. PMID 23050714
- [Background] List R, Gerber H, Foresti M, Rippstein P, Goldhahn J. A functional outcome study comparing total ankle arthroplasty (TAA) subjects with pain to subjects with absent level of pain by means of videofluoroscopy. Foot Ankle Surg. 2012 Dec;18(4):270-6. doi: 10.1016/j.fas.2012.04.001. Epub 2012 May 12. PMID 23093123
- [Background] Heller MO, Mehta M, Taylor WR, Kim DY, Speirs A, Duda GN, Perka C. Influence of prosthesis design and implantation technique on implant stresses after cementless revision THR. J Orthop Surg Res. 2011 May 13;6:20. doi: 10.1186/1749-799X-6-20. PMID 21569522
- [Background] Taylor WR, Kornaropoulos EI, Duda GN, Kratzenstein S, Ehrig RM, Arampatzis A, Heller MO. Repeatability and reproducibility of OSSCA, a functional approach for assessing the kinematics of the lower limb. Gait Posture. 2010 Jun;32(2):231-6. doi: 10.1016/j.gaitpost.2010.05.005. Epub 2010 May 23. PMID 20547061
- [Background] Stacoff A, Kramers-de Quervain IA, Luder G, List R, Stussi E. Ground reaction forces on stairs. Part II: knee implant patients versus normals. Gait Posture. 2007 Jun;26(1):48-58. doi: 10.1016/j.gaitpost.2006.07.015. Epub 2006 Sep 18. PMID 16979893
- See also: Institute of Biomechanics, ETH Zurich, Switzerland (Primary Study Site) — http://www.biomech.ethz.ch/
- See also: Free public database from instrumented implants, Charité - Universitätsmedizin Berlin Germany — http://www.orthoload.com/